CLINICAL TRIAL: NCT00917839
Title: Randomized, Placebo-Controlled Phase II Monocentric Trial for the Neuroprotective Effect of Lamotrigine Plus Interferon Beta 1a 30mcg Once Weekly Intramuscular in Patients With Relapsing-Remitting Multiple Sclerosis.
Brief Title: The Neuroprotective Effect of Lamotrigine and Interferon Beta 1a in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Dr. Norman Putzki, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LT.01
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: neuroprotection; multiple sclerosis; brain atrophy; mr-spectroscopy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lamotrigine (Experimental): 7 weeks initial phase with increasing dose beginning with 25 mg oral 12 months treatment phase with fixed dose of 100 mg oral
  Interventions: Drug: lamotrigine
- Placebo (Placebo Comparator): 300mg Mannitol with 2% Aerosil
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine — 100 mg, once daily, 12 months

SUMMARY:
This study is designed to evaluate the neuroprotective effect of lamotrigine in the combination of interferon beta 1a once weekly intramuscular in patients with relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* definitive multiple sclerosis according to Mc Donald criteria
* clinical isolated syndrome according to Mc Donald criteria
* Expanded Disability Status Scale Score 0-5
* Pre-treatment with interferon beta 1a (Avonex) since at least 2 months before inclusion

Exclusion Criteria:

* relapse within 30 days prior to randomisation
* steroid pulse therapy within 30 days prior to randomisation
* pregnancy or poor contraception
* contraindication for lamotrigine
* depressive symptoms
* drugs with possible interaction with lamotrigine according to instruction leaflet
* other medical relevant conditions but multiple sclerosis
* clinically relevant laboratory results
* contraindication for MRI
* missing informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
N-Acetyl-Aspartate / creatine - quotient in normal appearing white matter by MR-spectroscopy | 12 months
Safety of lamotrigine in combination with interferon beta 1a (30 mcg) once weekly intramuscular. | 6 months, 12 months

SECONDARY OUTCOMES:
relapse rate | 12 months
Expanded disability status score | 12 months
Fatigue Severity Score | 12 months
N-Acetyl-Aspartate / creatine - quotient in normal appearing white matter by MR-spectroscopy | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland